CLINICAL TRIAL: NCT06499740
Title: Adapting a Brief Suicide Intervention for Pediatric Primary Care: Enhancing Uptake and Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sarah Danzo, Assistant Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00019327; 1K23MH134229-01A1 (NIH)
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: It is anticipated that primary care physicians will deliver initial suicide risk screening, and will refer participating patients and their caregivers to an embedded social worker or integrated mental health clinician within the clinic who will deliver either treatment as usual (TAU; months 1 and 2 of the trial) or the pilot intervention (months 3 and 4 of the trial) to patients endorsing low to moderate suicide risk.
  Patients will only participate in treatment as usual or the pilot intervention. Outcomes will be compared across the TAU and intervention conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual (Active Comparator): Arm 1 entails months 1-2 of this study. Treatment as usual will be delivered by providers to adolescent patients in their clinics during the first two months of this study. Treatment as usual will be defined by each individual clinic based on their existing clinic protocols.
  Interventions: Behavioral: Treatment as Usual
- SAFETY-A Based Adapted Intervention (Experimental): Arm 2 entails months 3-4 of this study. Participating providers will deliver the adapted intervention for the second half (months 3-4) of the pilot trial. The intervention will be based on the evidence-based SAFETY-Acute protocol and will be adapted based on information from potential users prior to piloting. It is anticipated that both adolescent patients and their parents/caregivers will be involved in the intervention. Anticipated components of the intervention include safety planning, lethal means restriction, communication, identifying adolescent and family strengths, and linking to longer term care.
  Interventions: Behavioral: Adapted SAFETY-A for PC

INTERVENTIONS:
Behavioral: Adapted SAFETY-A for PC — This intervention is a suicide prevention intervention that will be adapted from the evidence-based SAFETY-Acute program. The specific intervention components will be determined from information gathered in this study but the investigators anticipate will include components such as safety planning, lethal means restriction, psychoeducation, motivation building, and care linkage.
  Arms: SAFETY-A Based Adapted Intervention
Behavioral: Treatment as Usual — Treatment as usual delivered in participating clinics.
  Arms: Treatment as usual

SUMMARY:
Suicide is a leading cause of death among adolescents in the United States and improving access to high quality just-in-time suicide interventions to reduce risk has important public health implications. Integrating such interventions into routinely accessed settings, such as pediatric primary care, holds promise; however, many clinicians in these settings fail to adequately screen or intervene in youth suicidal thoughts and behaviors, representing a key barrier to reducing suicide. The proposed study is a pre-post quasi-experimental pilot feasibility and preliminary efficacy trial of an adaptation of the SAFETY-Acute suicide prevention intervention implemented in 3 pediatric primary care clinics.

DETAILED DESCRIPTION:
This project aims to take an innovative, user-centered design approach to adapt and optimize a brief, evidence-based suicide intervention, SAFETY-Acute (SAFETY-A; formerly known as Family Intervention for Suicide Prevention -aka FISP), for use in primary care settings to support primary care management of adolescents with low to moderate risk suicidal thoughts and behaviors (STB). In this trial, the investigators will conduct a pre-post quasi-experimental pilot feasibility and preliminary efficacy trial of an adapted STB model of care based of the SAFETY-Acute intervention, compared to treatment as usual, with 3 primary care clinics. The trial will include 48 10-18-year-old patients with STB and their parents/caregivers (16 dyads per clinic). The investigators will assess acceptability and feasibility of the STB model of care, preliminary intervention impacts, and need for further adaptation.

ELIGIBILITY:
Inclusion Criteria:

* adolescent between the ages of 10 and 18 years old
* speaks fluent English
* current or past low to moderate suicide risk (denies current plan or intent to kill self)

Exclusion Criteria:

* high suicide risk (endorses current plan or intent or ASQ score =5, or prior attempt within last 3 months)
* does not speak fluent English

Note: Caregivers of 10-18 yr olds will also be included so age limits for participating samples include:

1. Adolescents: ages 10-18 years old
2. Parents/Caregivers: ages 18 years and older

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | Participant and providers complete approximately 2 weeks after completing intervention
  Feasibility of the intervention (includes 4 items scored on a 5 point likert scale with higher scores representing greater feasibility.)
Acceptability of Intervention Measure | Participant and providers complete approximately 2 weeks after completing intervention
  Participant rated acceptability of the intervention (includes 4 items scored on a 5 point likert scale with higher scores representing greater acceptability.)
Intervention Appropriateness Measure | Participant and providers complete approximately 2 weeks after completing intervention
  Participant rated appropriateness of the intervention (includes 4 items scored on a 5 point likert scale with higher scores representing greater appropriateness.)
Client Satisfaction Questionnaire | Participant completes approximately 2 weeks after completing intervention
  Caregiver participant rated satisfaction with the intervention (includes 8 items scored on a 4 point likert scale with higher scores representing greater satisfaction.)
Youth Satisfaction Questionnaire | Participant completes approximately 2 weeks after completing intervention
  Adolescent participant rated satisfaction with the intervention (includes 5 items scored on a 3 point likert scale with higher scores representing greater satisfaction.)
Intervention Usability Scale | Participant/provider completes approximately 2 weeks after completing intervention
  Participant rated intervention usability (includes 10 items scored on a 5 point likert scale with greater total score representing greater usability).

SECONDARY OUTCOMES:
Parent Self Efficacy Scale | Participant completes at baseline, approximately 2 weeks after completing intervention, and again 2 months following the intervention
  Caregiver rated self-efficacy of being able to keep youth safe (includes 5 items scored on a 5 point likert scale with greater total score representing greater parent self-efficacy).
Adapted General Self-Efficacy Scale | Participant completes at baseline, approximately 2 weeks after completing intervention, and again 2 months following the intervention
  Patient rated self-efficacy of being able to keep self safe (includes 10 items scored on a 4 point likert scale with greater total score representing greater self-efficacy).
adapted Child Parent Relationship Scale | Participant completes at baseline, approximately 2 weeks after completing intervention, and again 2 months following the intervention
  Patient and caregiver rated family involvement/relationship quality (includes 15 items scored on a 5 point likert scale with two subscales [closeness and conflict] where higher total score on each subscale represents greater closeness or conflict).

OTHER OUTCOMES:
Ask Suicide Screening Questions (ASQ) | Participant completes at baseline, approximately 2 weeks after completing intervention, and again 2 months following the intervention
  Exploratory suicide and mental health outcomes (includes 5 items scored as yes/no with greater number of yes or a yes on item 5 representing greater suicide risk).
Revised Children's Anxiety and Depression Scale-25 | Participant completes at baseline, approximately 2 weeks after completing intervention, and again 2 months following the intervention
  Exploratory suicide and mental health outcomes (includes 25 items scored on a 4 point likert scale with higher total score representing greater symptom severity).
Diagnostic and Statistical Manual of Mental Disorders-5 cross cutting assessment | Participant completes at baseline, approximately 2 weeks after completing intervention, and again 2 months following the intervention
  Exploratory suicide and mental health outcomes (includes 25 items scored on a 4 point likert scale with higher scores representing greater symptom severity).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Danzo, PhD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No
Plan is currently undecided and will be updated prior to clinical trial beginning.